CLINICAL TRIAL: NCT06628466
Title: Clinical Response of Nuberol Forte in Chronic Neck Pain in Routine Rehabilitation Centers
Acronym: "NOTICE"
Status: Completed | Type: Observational
Sponsor: The Searle Company Limited Pakistan (Industry)
Responsible Party: Sponsor
Other Study IDs: TSCL-NOTICE_001
Record Dates: First submitted 2024-03-19; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-03

CONDITIONS: Chronic Neck Pain
Keywords: Chronic Neck Pain; Paracetamol Orphenadrine combination; Physiotherapy; Pakistan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients of either sex between the ages 18 and 70 years, suffering from Chronic neck pain: Each patient will begin with the start of physical therapy with Nuberol Forte for the symptomatic management of the chronic neck pain. Subjects will be observed for overall safety and effectiveness of study drug from visit 1 (baseline visit, screening and start of treatment), to visit 2 (Week 1-2, end of treatment) in the routine practice.
  Interventions: Drug: Nuberol Forte

INTERVENTIONS:
Drug: Nuberol Forte — Quality of Life study

SUMMARY:
Globally, the prevalence of neck pain ranges from 16.7% to 75.1%. Despite conducting multiple studies on specific subject pools in Pakistan, primarily focusing on professional-related neck pain, there is a lack of accurate data to determine the local prevalence of neck pain or the effective management of neck pain through physical therapy and pharmacological intervention. The purpose of this study is to evaluate the clinical effectiveness of paracetamol and orphenadrine (Nuberol Forte) when combined with physical therapy in Pakistani patients suffering from neck pain at regular rehabilitation centers.

DETAILED DESCRIPTION:
For most cases of neck pain, the risk factors are multifactorial, and clear pathophysiological mechanisms are lacking. Treatment efforts aim to alleviate symptoms in the absence of causal treatment alternatives, while rehabilitation programs enhance the functional status. Therefore, it is imperative to have validated questionnaires to measure pain, other symptoms, and functional limitations in neck pain disorders, both for characterizing the patient group and evaluating rehabilitation efforts. The Alfta Rehab Center developed the Profile Fitness Mapping for Neck (ProFitMap-neck) questionnaire between 1992 and 1994, which comprises two scales for assessing self-estimated symptoms and functional limitations resulting from neck problems. The symptom scale comprises two indices, representing the intensity and frequency of the symptoms, while the functional limitation scale produces a single function index. The current study describes and evaluates the reliability and validity of a Profile Fitness Mapping Neck questionnaire (ProFitMap-neck) to assess the symptoms and functional limitations of Pakistani people with chronic neck pain. There is no clear evidence that orphenadrine's antimuscarinic activity is related to its antinociceptive action, although its mild antihistaminic activity may play a role. Histamine can stimulate nociceptors, and histamine receptors are found in brain tissue and primary afferent neurons. Unlike the other muscle relaxants, orphenadrine produces some independent analgesic effects that may contribute to its efficacy in relieving painful skeletal muscle spasm. Paracetamol/acetaminophen is one of the most popular and commonly used analgesic and antipyretic drugs in the world, available without a prescription in both mono- and multi-component preparations. Patients who cannot receive treatment from non-steroidal anti-inflammatory drugs (NSAIDs), such as those with bronchial asthma, peptic ulcer disease, hemophilia, salicylate-sensitized individuals, or pregnant or breastfeeding women, opt for this drug. The mechanism of action is complex and includes the effects of both the peripheral (COX inhibition) and central (COX, serotonergic descending neuronal pathway, L-arginine/NO pathway, cannabinoid system) antinociception processes, as well as redox mechanisms that block the production of chemicals in the body that are responsible for pain. Paracetamol is a well-tolerated drug and produces few side effects from the gastrointestinal tract. The non-clinical data demonstrated that orphenadrine is a mild antinociceptive agent similar to non-opioid analgesics. There are clear indications that the combination with Paracetamol may provide increased antinociceptive activity and duration of action over and above Orphenadrine or Paracetamol alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a clinical history of chronic neck pain from last 3 months.
* Patient aged ≥18 and ≤70 years inclusive of either sex.
* Patient with ability to understand and sign written informed consent form.

Exclusion Criteria:

* Subjects with acute or subacute neck pain.
* Subjects with specific etiology for neck pain (e.g. trauma, herniated disc, vertebral deformities, fractures);
* Subjects with central or peripheral neurological signs.
* Individuals with systemic diseases, neuromuscular diseases, rheumatic diseases, cognitive deficit, tumors.
* Known hypersensitivity to Nuberol Forte product, the metabolites, or formulation excipients.
* Patients with Glaucoma, prostatic hypertrophy or obstruction at the bladder neck, myasthenia gravis, oesophageal spasm and pyloric or duodenal obstruction.
* Treated with Nuberol Forte to evaluate safety as per approved prescribing information for Nuberol Forte in Pakistan.
* Pregnant (assesed on LMP) or breast feeding women (assessed on interview).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population including patients of either sex between the ages 18 and 70 years, suffering from Neck pain, will be enrolled in the study in random order. The random number will be marked using a random number table. In each case, before recruitment, the subject pain intensity measures the Numerical Rating Scale (NRS) for pain.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
To assess the improvement in the symptoms and functional limitations of chronic neck pain by physical therapy along with Nuberol Fort (paracetamol orphenadrine combination). | From baseline to week 2
  The questionnaire Profile Fitness Mapping for neck (ProFitMap-neck) consists of two scales designed for the assessment of self-estimated symptoms and functional limitations due to neck problems. The symptom scale consists of two indices of separate aspects of symptomatology, the intensity and the frequency of the symptoms, and the functional limitation scale yields one function index. The calculated score for very often from 1-6, 1 score never (minimum) and 6 score often (maximum). The score 7-12 for how much, 7 score nothing (Better) and 12 score unbearable (Worst)
To assess the change of improvement in pain intensity, the pain intensity assesses by NRS scale. | From baseline to week 2
  Pain intensity assess by Numeric Pain Rating Scale (NRS). The pain score 0, no pain (Minimum) and 10, severe pain (Maximum).
  0 (no pain), 1-3 (Mild Pain), 3-7 (moderate Pain), 7-10 (severe pain), 10 & above (worst Pain)

SECONDARY OUTCOMES:
To assess The overall safety of Paracetamol orphenadrine combination in chronic neck pain. | From baseline to week 2
  Safety of Nuberol Forte (Paracetamol Orphenadrine combination) will assess based on the incidence of reported TEAEs by system organ class ; preferred term, as well as by categories: TEAE, severe TEAE, serious TEAE, drug-related TEAE, drug-related severe TEAE, drug-related serious TEAE, TEAE leading to discontinuation, ; TEAE with outcome of death. Drug-related TEAEs were defined as TEAEs assigned a Study Drug (Nuberol Forte) relationship of adverse reaction; suspected adverse reaction. TEAEs were coded using the Medical Dictionary for Regulatory Activities, version 19.0. The severity of TEAEs are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03. TEAEs were defined as any adverse event that started or increased in severity after the first dose of Study Drug on Day 1 through the Final Study Visit (2 weeks +/-3 days after last dose).

CONTACTS AND LOCATIONS:
Overall Officials: Zahoor Ahmed, Neurologist, Principal Investigator — Karachi medical Complex, Karachi; Ali Hassan, Neurologist, Principal Investigator — Ziauddin Hospital, Karachi; Sonober Jawaid, Neurologist, Principal Investigator — Al-Maisarah Hospital, Karachi; Muhammad Y Ahmedani, FCPS, Principal Investigator — Baqai Hospital, Karachi; Ghufranullah Khan, Surgeon, Principal Investigator — Tabba Heart, Karachi; Jai S Rana, Neurologist, Principal Investigator — Poly Medical & Dental Clinic, Karachi
Locations (1):
- The Searle Company Limited, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjorklund M, Hamberg J, Heiden M, Barnekow-Bergkvist M. The assessment of symptoms and functional limitations in low back pain patients: validity and reliability of a new questionnaire. Eur Spine J. 2007 Nov;16(11):1799-811. doi: 10.1007/s00586-007-0405-z. Epub 2007 Jun 22. PMID 17587068
- [Background] Young IA, Dunning J, Butts R, Cleland JA, Fernandez-de-Las-Penas C. Psychometric properties of the Numeric Pain Rating Scale and Neck Disability Index in patients with cervicogenic headache. Cephalalgia. 2019 Jan;39(1):44-51. doi: 10.1177/0333102418772584. Epub 2018 Apr 19. PMID 29673262
- [Background] Thong ISK, Jensen MP, Miro J, Tan G. The validity of pain intensity measures: what do the NRS, VAS, VRS, and FPS-R measure? Scand J Pain. 2018 Jan 26;18(1):99-107. doi: 10.1515/sjpain-2018-0012. PMID 29794282
- [Background] Hunskaar S, Donnell D. Clinical and pharmacological review of the efficacy of orphenadrine and its combination with paracetamol in painful conditions. J Int Med Res. 1991 Mar-Apr;19(2):71-87. doi: 10.1177/030006059101900201. PMID 1864455
- [Background] McGuinness BW. A double-blind comparison in general practice of a combination tablet containing orphenadrine citrate and paracetamol ('Norgesic') with paracetamol alone. J Int Med Res. 1983;11(1):42-5. doi: 10.1177/030006058301100109. PMID 6219903
- [Background] Hoivik HO, Moe N. Effect of a combination of orphenadrine/paracetamol tablets ('Norgesic') on myalgia: a double-blind comparison with placebo in general practice. Curr Med Res Opin. 1983;8(8):531-5. doi: 10.1185/03007998309109793. PMID 6653131
- [Background] Straube A, Aicher B, Fiebich BL, Haag G. Combined analgesics in (headache) pain therapy: shotgun approach or precise multi-target therapeutics? BMC Neurol. 2011 Mar 31;11:43. doi: 10.1186/1471-2377-11-43. PMID 21453539
- [Background] Bogduk N. The anatomy and pathophysiology of neck pain. Phys Med Rehabil Clin N Am. 2011 Aug;22(3):367-82, vii. doi: 10.1016/j.pmr.2011.03.008. PMID 21824580
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Alsultan F, De Nunzio AM, Rushton A, Heneghan NR, Falla D. Variability of neck and trunk movement during single- and dual-task gait in people with chronic neck pain. Clin Biomech (Bristol). 2020 Feb;72:31-36. doi: 10.1016/j.clinbiomech.2019.11.019. Epub 2019 Nov 28. PMID 31809920
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Palazzo C, Ravaud JF, Papelard A, Ravaud P, Poiraudeau S. The burden of musculoskeletal conditions. PLoS One. 2014 Mar 4;9(3):e90633. doi: 10.1371/journal.pone.0090633. eCollection 2014. PMID 24595187
- [Background] Duffield SJ, Ellis BM, Goodson N, Walker-Bone K, Conaghan PG, Margham T, Loftis T. The contribution of musculoskeletal disorders in multimorbidity: Implications for practice and policy. Best Pract Res Clin Rheumatol. 2017 Apr;31(2):129-144. doi: 10.1016/j.berh.2017.09.004. Epub 2017 Nov 1. PMID 29224692